CLINICAL TRIAL: NCT02672358
Title: A Phase II, Multi-center, Single Arm, Open Label Study to Assess Efficacy and Safety of Dabrafenib and Trametinib Combination Therapy in Japanese Patients With BRAF V600E Mutation Positive Metastatic (Stage IV) Non-small Cell Lung Cancer
Brief Title: Study of Efficacy and Safety of Dabrafenib and Trametinib Combination Therapy in Japanese Patients With BRAF V600E Stage IV NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDRB436E1201
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; NSCLC; dabrafenib; trametinib; Japanese patients; BRAF V600E mutation positive metastatic; stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib +Trametinib (Experimental): Oral Dabrafenib plus Oral Trametinib
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Oral Dabrafenib 150 mg BID
Drug: Trametinib — Oral Trametinib 2 mg QD

SUMMARY:
This is an open-label, multicenter, non-randomized, single arm, phase II study to assess efficacy and safety of the dabrafenib and trametinib combination in Japanese patients with any line, stage IV NSCLC harboring a confirmed BRAF V600E mutation.

Patients will receive oral dabrafenib twice daily and oral trametinib once daily combination therapy. Patients may continue study treatment until disease progression, unacceptable adverse events, start of a new anti-cancer therapy, consent withdrawal, death, or end of the study. Patients who have met the criteria for disease progression (PD) according to RECIST v1.1 may continue to receive study treatment if the investigator believes the patient is receiving clinical benefit and the patient is willing to continue on study treatment. After discontinuation of study treatment, all patients will be followed for survival until death, lost to follow-up, withdrawal of consent, or end of study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of NSCLC stage IV (according to AJCC Staging 7th Edition)
* Presence of a BRAF V600E mutation in lung cancer tissue. BRAF V600E mutation tested by local laboratory (e.g. study center laboratory, local laboratory company) with proper quality control and license to operation by local health authority is allowed.
* Measurable disease according to RECIST v1.1.

Exclusion Criteria:

* Previous treatment with a BRAF inhibitor (including but not limited to dabrafenib, vemurafenib, encorafenib, and XL281/BMS-908662) or MEK inhibitor (including but not limited to trametinib, cobimetinib, binimetinib, AZD6244, and RDEA119) prior to start of study treatment
* Patients with brain metastases are excluded if their brain metastases are:

  * Symptomatic OR
  * Treated (surgery, radiation therapy) but not clinically and radiographically stable 3 weeks after local therapy (as assessed by contrast enhanced magnetic resonance imaging [MRI] or computed tomography [CT]), OR
  * Asymptomatic and untreated but >1 cm in the longest dimension
* History of malignancy with confirmed activating RAS mutation at any time.
* History of interstitial lung disease or pneumonitis
* A history or current evidence of retinal vein occlusion (RVO)
* Current evidence of unstable aneurysm or one that needs treatment

Other protocol-defined inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-03 (Estimated); Primary Completion 2019-09-02 (Estimated); Study Completion 2020-12-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by investigator assessment | Approximately 2 years
  ORR, defined as the percentage of patients with a confirmed CR or PR by investigator assessment as per RECIST v1.1 criteria

SECONDARY OUTCOMES:
Duration of response (DOR) | Approximately 2 years
  DOR, defined for the subset of patients with confirmed CR or PR, as the time from first documented evidence of CR or PR until time of first documented disease progression or death due to any cause.
Disease control rate (DCR) | Approximately 2 years
  DCR, defined as the proportion of patients with best overall response of CR, PR, or SD.
Progression-free survival (PFS) | Approximately 2 years
  PFS, defined as the interval between first dose and the earliest date of disease progression or death due to any cause.
Overall survival (OS) | Approximately 2 years
  OS, defined as the time from the date of first dose until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com